CLINICAL TRIAL: NCT06061549
Title: A Phase 1b, Pilot Trial Evaluating the Safety and Pharmacodynamic Effects of SRD-001 (AAV1-SERCA2a) in Subjects With Heart Failure With Preserved Ejection Fraction
Brief Title: Modulation of SERCA2a of Intra-myocytic Calcium Trafficking in Heart Failure With Preserved Ejection Fraction
Acronym: MUSIC-HFpEF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sardocor Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRD-001-1003
Record Dates: First submitted 2023-07-30; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure, Diastolic; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRD-001 Gene Therapy (Experimental): AAV1/SERCA2a 3E13 vg
  Interventions: Biological: AAV1/SERCA2a

INTERVENTIONS:
Biological: AAV1/SERCA2a — 3E13 viral genomes fixed dose

SUMMARY:
The goal of this clinical trial is to test an experimental gene therapy in participants with heart failure with preserved ejection fraction, also known as diastolic heart failure. The main questions it aims to answer are:

* safety and tolerability of the gene therapy; and
* whether the gene therapy helps the heart ventricles relax during filling. Participants will undergo a one-time infusion of the gene therapy in the cardiac catheterization laboratory and then be followed for safety and effects on left-sided filling pressures while exercising. The first year will have multiple in-person visits followed by 4 years of biannual phone calls.

DETAILED DESCRIPTION:
Eligible participants will undergo a one-time antegrade epicardial coronary artery infusion of gene therapy delivered to the 3 major cardiac territories of the left ventricle of the heart (anterior, lateral, inferior/posterior) or bypass grafts unless contraindicated. Post-procedure, the subject will be monitored continuously for a minimum of 4 hours and then discharged to home that same day if medically appropriate. Participants will be followed for 52 weeks as part of the main trial. On Day 2 and Week 1, subjects will be contacted by phone for a general safety assessment, and if clinically indicated, an in-person evaluation and assessment will be performed as soon as possible. On Weeks 2, 4, 12, 24 and 52, subjects will undergo general safety assessments. Additionally, at Weeks 24 and 52, subjects will undergo outpatient core resting and exercise transthoracic echocardiography, right heart catheterization with hemodynamic monitoring and gas exchange measurements, 6-minute wall test, cardiac biomarker testing and completion the Kansas City Cardiomyopathy Questionnaire. Upon completion of the active observation period, participants will continue to be followed for 4 years with bi-annual, semi-structured telephone or in-person questionnaires that collect information on overall status and other comorbid conditions of interest in gene therapy trials.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Negative for anti-AAV1 neutralizing antibodies
* NYHA class II or III
* Left ventricular ejection fraction ≥ 50%
* Evidence of resting or exercise-induced left ventricle filling pressure
* On oral diuretic therapy
* Adequate birth control

Exclusion Criteria:

* NYHA class IV
* Heart failure requiring hospitalization in the past 3 months
* Manifested or provocable ischemic heart disease
* Atrial fibrillation
* History of congenital heart disease, restrictive or infiltrative cardiomyopathy, hypertrophic cardiomyopathy, acute myocarditis, pericardial disease, uncorrected thyroid disease or discrete left ventricular (LV) aneurysm
* History of amyloidosis
* Untreated left-sided valvular disease
* Severe COPD
* BMI > 50 kg/m^2
* Severe liver, kidney or hematologic dysfunction
* Cancer within the past 5 years
* Unstable concurrent conditions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary capillary wedge pressure (PCWP) | Week 24 and Week 52
  PCWP assessed by right heart catheterization; change in mmHg from baseline

SECONDARY OUTCOMES:
Change in PCWP at 20W exercise | Week 24 and Week 52
  PCWP assessed by right heart catheterization; change in mmHg from baseline
Change in oxygen uptake (VO2) during exercise | Week 24 and Week 52
  VO2 assessed by bicycle exercise; change in mL/min from baseline
Change in left ventricular (LV) relaxation | Week 24 and Week 52
  Assessed by transesophageal echocardiography (ultrasound) using 2 methods: LV global peak early diastolic strain rate (1/s) and LV tau
Change in NT-proBNP | Week 24 and Week 52
  Laboratory measurement (picograms per mL) in blood; high levels indicate the heart is working too hard to pump blood; decrease over time would indicate an improvement in heart failure condition
Change in left atrial end systolic volume | Week 24 and Week 52
  Assessed by transesophageal echocardiography (ultrasound); change in mL/m2 from baseline
Change in left atrial reservoir strain | Week 24 and Week 52
  Assessed by transesophageal echocardiography (ultrasound); change in %from baseline
Change in left atrial contractile strain | Week 24 and Week 52
  Assessed by transesophageal echocardiography (ultrasound); change in % from baseline
Change in 6 Minute Walk Distance | Week 24 and Week 52
  Distance walked in 6 minutes, measured in meters; the longer distance walked, the better medical condition
Change in 6 Minute Walk Test Borg scale | Week 24 and Week 52
  Self-rated shortness of breath score with scale from 0 to 10, ranging from none to very, very severe
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | Week 24 and Week 52
  Measures symptoms, physical and social limitations, and quality of life in patients with heart failure; 23-item self-administered questionnaire; score of 0 to 100; 0-24, very poor to poor; 25-49, poor to fair; 50 to 74, faire to good; and 75 to 100, good to excellent
Change in New York Heart Association class | Week 24 and Week 52
  Classification of heart failure based on severity of symptoms; 4 classes, I, II, III or IV where class I is having no symptoms doing ordinary physical activity; class II is having fatigue, shortness of breath, palpitations or angina with ordinary physical activity; class II is being comfortable only at rest; and class IV is having symptoms even at rest

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No